CLINICAL TRIAL: NCT07340034
Title: Effects of Focal Muscle Vibration Versus Whole Upper Limb Vibration on Spasticity and Upper Motor Control Functions in Post-Stroke Patients
Brief Title: Effects of Focal Muscle Vibration Versus Whole Upper Limb Vibration in Post-Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/036
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Post Stroke Upper Limb Spasticity
Keywords: Whole upper limb vibration; Focal muscle vibration; Upper limb spasticity; Upper Motor Control Functions
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This study will use a parallel-group design, with participants randomly allocated into two intervention groups.
  Group A (Focused Muscle Vibration - FMV) 30-minute session: 15 min upper-extremity ROM/stretching + 15 min FMV. FMV delivered at 30 Hz while seated (shoulder slightly abducted, elbow at 90°). Vibration applied in 60-s bouts with 60-s rest. Target muscles: biceps, triceps, anterior deltoid, FDS, FCR, ECR, ECU.
  Frequency: 5 days/week for 8 weeks. Group B (Upper Limb Vibration ULV) 30-minute session: 15 min ROM/stretching + ULV using Power Plate Pro5. Seated position with elbow 70-80° flexion and wrist dorsiflexed. ULV applied in 2 × 60-s bouts, 1-min rest, amplitude 2 mm, frequency 35-40 Hz.
  Frequency: 5 days/week for 8 weeks. Participants will be randomly allocated into two parallel groups to ensure an unbiased comparison, with each group receiving its specific intervention protocol throughout the study period without crossover to the other groups intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: outcome assessor will be blind about participants allocation; this will ensure that their evaluations are objective and not influenced by knowledge of which treatment group participants belong to. Participants in both groups will be masked to the treatment of the other group by scheduling their sessions at different times
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focal muscle vibration through focal muscle vibrator along with conventional neurorehabilitation (Experimental): Group A will receive the Focal muscle vibration in the major group of muscle such as Elbow flexors and wrist flexors along with the conventional neurorehabilitation.
  Interventions: Other: Focal muscle vibration through focal muscle vibrator along with conventional neurorehabilitation
- Upper limb vibration through whole body vibrator along with conventional neurorehabilitation (Active Comparator): Group B will receive the upper limb vibration which will include all muscles of effected limb along with the conventional neurorehabilitation.
  Interventions: Other: Upper limb vibration through whole body vibrator along with conventional neurorehabilitation

INTERVENTIONS:
Other: Focal muscle vibration through focal muscle vibrator along with conventional neurorehabilitation — Group A will receive the 30 minutes treatment protocol. Warm-up exercises for first 15 minutes with ROM and stretching exercises of upper extremity 15 minutes application of FMV All participants were instructed to sit back in a high, fixed chair without armrests, keeping their feet flat on the floor. The dominant shoulder was positioned slightly away from the trunk i.e. in slight abduction and the elbow was held at a 90° angle as part of the designated vibration position. After setting up, the researcher guided the participants to remain seated in the same position as it might affect the results and treatment. The participants then received the vibration in frequency of 30 Hz in both vertical and horizontal directions.
  Based on our review of prior clinical studies aimed at improving muscle spasticity we implemented vibration protocols with exposure times ranging from 30 to 60 seconds and rest intervals between 15 and 60 seconds. The analysis focused on seven muscle groups
  Arms: Focal muscle vibration through focal muscle vibrator along with conventional neurorehabilitation
Other: Upper limb vibration through whole body vibrator along with conventional neurorehabilitation — Group B will receive the 30 minutes treatment protocol. Warm-up exercises for first 15 minutes with ROM and stretching exercises of upper extremity.
  Patients in the treatment group received upper limb vibration using the Power Plate vibration platform (Performance Health Systems, Power Plate Pro5, North America 2009). The patient was seated on a stool placed next to the whole-body vibration device; the elbow was positioned at 70-80 degrees flexion and wrist was positioned at dorsiflexion and upper limb vibration was applied through Whole body vibrator to the affected limb for two minutes. The WBV consisted of two sessions of 60 seconds of stimulation interrupted by a one-minute break between each session to prevent muscle fatigue. The amplitude of the vibration was 2 mm, and the frequency was 35-40 Hz. An experienced physical therapist supervised the WBV administration. The upper limb vibration treatment was performed 5 times a week for 8 weeks.
  Arms: Upper limb vibration through whole body vibrator along with conventional neurorehabilitation

SUMMARY:
This study contributes to the growing body of knowledge on rehabilitation strategies for post-stroke patients, specifically focusing on the efficacy of vibration therapy modalities. By comparing focal muscle vibration therapy and whole upper limb vibration therapy, the research aims to provide empirical evidence that can inform clinical practices and enhance rehabilitation outcomes. The findings are expected to clarify which modality is more effective in reducing spasticity and improving motor control, thereby guiding clinicians in selecting appropriate interventions tailored to individual patient needs, increasing chances of benefits, time management and useful for academic purpose. Furthermore, the study addresses a critical gap in the literature, facilitating further research and discussion on the mechanisms underlying vibration therapy's effects.

Ultimately, this research aims to reduce spasticity and improve community outcomes by enhancing the quality of life for stroke survivors, enabling them to regain independence and participate more fully in daily activities by regaining the motor control functions. By contributing to both theoretical and practical frameworks, the study seeks to advance the field of neurorehabilitation and support informed decision-making among healthcare professionals.

DETAILED DESCRIPTION:
Motor impairment post-stroke, which usually affects the movement of the face, arm, and leg on one side of the body, impacts approximately 80% of individuals who have experienced a stroke. Upper limb motor impairments (involving the arm, hand, and/or fingers) are often long-lasting and debilitating; only about half of stroke survivors with an initially paralyzed upper limb recover some useful function within six months.

Recently, mechanical vibrations have been utilized as a form of somatosensory stimulation to enhance motor function and to address muscle spasticity in the upper limbs following a stroke. When applying vibration stimuli during exercise or physical rehabilitation, these can be broadly classified into two categories: (a) vibrations that are directly applied to a specific muscle or tendon, and (b) indirect vibrations that are not limited to a specific muscle, delivered either through the feet while standing on a platform or through the hands using a handheld device. The direct application of vibrations to a muscle or tendon is often referred to as focal muscle vibration (FMV) or segmental vibration (SV), and it may also be called repetitive muscle vibration (rMV). In contrast, indirect vibrations delivered through the hands are typically known as upper limb vibration (ULV), while those aimed at the lower limbs are referred to as whole-body vibration (WBV).

Vibration therapy (VT) is a form of physical therapy that employs mechanical vibration waves to stimulate the human neuromuscular system for therapeutic benefits. It demonstrates promising potential for use in the rehabilitation of dysfunctions part of bosy resulting from a stroke.

Focal muscle vibration (FMV) OR segmental muscle vibration is a relatively new approach used to enhance motor function and reduce spasticity in the hemiplegic upper limb of stroke patients. In FMV, a vibratory stimulus is delivered to a specific muscle tendon via a mechanical device, which activates the muscle spindle primary endings and generates Ia inputs. Vibration applied to a muscle can elevate the motor-evoked potential recorded from that muscle at rest, indicating an increase in corticospinal excitability during the vibration. Additionally, studies have shown that the duration of the cortical silent period in a forearm flexor muscle can increase when the antagonist forearm extensors are vibrated, providing strong evidence that pure sensory stimulation can influence motor cortical excitability.

ELIGIBILITY:
INCLUSION CRITERIA Clinical diagnosis of first-ever ischemic stroke Age from 45 to 60 years Both male and female participants Onset of stroke 3 month to 6 months previously Modified Ashworth Scale (MAS) score for the upper limb muscles on the hemiparetic side between 1+ and 3 Able to follow verbal commands and sign informed consent forms EXCLUSION CRITERIA Cardiovascular disease or uncontrolled diabetes Upper limb muscle contracture on the affected side Peripheral neuropathy Uncontrolled hypertension Malignant tumors Uncontrolled seizures Dementia

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer assessment of upper limb (FMA-UE) | baseline, after 2 weeks and 4 weeks
  The Fugl-Meyer Assessment-Upper Extremity (FMA-UE) is a commonly utilized tool for measuring motor impairment in stroke rehabilitation. The FMA-UE has demonstrated excellent test-retest and inter- and intra-rater reliability, and evidence for its content validity in acute and subacute populations have been widely reported. The UE section of the FMA consists of 33 items and is scored on a 3-point ordinal scale with 0 meaning cannot perform, 1 meaning can partially perform, and 2 meaning can perform fully. Scores are summed with a maximum potential score of 66 points.
Modified Ashworth scale (MAS) | baseline, after 4 weeks and 8 weeks
  The Modified Ashworth Scale (MAS) is the most widely used clinical tool for measuring increased muscle tone or spasticity The MAS has demonstrated excellent test-retest and inter- and intra-rater reliability, The inter-rater reliability of the scale has been reported to vary significantly depending on the muscle group being assessed, the examiner's experience, and methodological inconsistencies in applying the scale.
  The scale is as follows:
  0: No increase in muscle tone
  1. Slight increase in muscle tone, with a catch and release or minimal resistance at the end of the range of motion when an affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested as a catch, followed by minimal resistance through the remainder (less than half) of the range of motion
  2. A marked increase in muscle tone throughout most of the range of motion
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu YH, Chen HJ, Liao CD, Chen PJ, Wang XM, Yu CH, Chen PY, Lin CH. Upper extremity function and disability recovery with vibration therapy after stroke: a systematic review and meta-analysis of RCTs. J Neuroeng Rehabil. 2024 Dec 21;21(1):221. doi: 10.1186/s12984-024-01515-6. PMID 39707380
- [Background] Karnath HO. Pusher syndrome--a frequent but little-known disturbance of body orientation perception. J Neurol. 2007 Apr;254(4):415-24. doi: 10.1007/s00415-006-0341-6. Epub 2007 Mar 25. PMID 17385082